CLINICAL TRIAL: NCT00523744
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Tolerability of a 4 Week Therapy With the Fixed Dose Combination of Amlodipine 10 mg Plus Valsartan 160 mg in Hypertensive Patients Not Adequately Responding to a 4 Week Therapy With the Free Combination of an Angiotensin Receptor Blocker (Olmesartan 20 mg) Plus Amlodipine 10 mg
Brief Title: Efficacy and Safety of Valsartan and Amlodipine (± HCTZ) in Adults With Moderate, Inadequately Controlled Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489ADE06
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
Keywords: hypertension, valsartan, amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Olmesartan Medoxomil; Amlodipine, Valsartan Drug Combination; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amlodipine(AML)+olmesartan, AML+valsartan, AML+valsartan+HCTZ (Experimental): During the Treatment Phase 1, participants received 1 week of treatment with olmesartan 10 mg and amlodipine 5 mg once daily in free combination, followed by three weeks of treatment with olmesartan 20 mg plus amlodipine 10 mg once daily in free combination. During the treatment Phase 2 of the study participants received amlodipine 10 mg plus valsartan 160 mg for 4 weeks. During the Extension Phase, participants received 4 weeks treatment with amlodipine 10 mg plus valsartan 160 mg plus hydrochlorothiazide (HCTZ) 12.5 mg.
  Interventions: Drug: Amlodipine; Drug: Olmesartan medoxomil; Drug: Amlodipine+valsartan; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Amlodipine — Amlodipine supplied as 5 mg tablets, taken orally once a day during Treatment Phase 1 only.
Drug: Olmesartan medoxomil — Olmesartan medoxomil supplied as 10 mg tablets taken once a day during Treatment Phase 1 only.
Drug: Amlodipine+valsartan — Fixed-dose combination of amlodipine 10 mg plus valsartan 160 mg tablet taken orally once a day during Treatment Phase 2 and Extension Phase.
  Other Names: Exforge
Drug: Hydrochlorothiazide — Hydrochlorothiazide (HCTZ) 12.5 mg tablets taken once a day during the Extension Phase.
  Other Names: Sandoz

SUMMARY:
This study will evaluate the efficacy and safety of valsartan and amlodipine in fixed dose combination in adults with moderate, inadequately controlled hypertension. There was an optional study extension for eligible patients who wanted to participate that contains the triple therapy (ie, hydrochlorothiazide+ amlodipine/valsartan).

DETAILED DESCRIPTION:
Title of study extension: An open-label, multicenter extension to evaluate the efficacy and tolerability of a 4 week therapy with hydrochlorothiazide 12.5 mg plus amlodipine 10 mg/valsartan 160 mg in hypertensive patients not adequately responding to a 4 week therapy each with the combinations of olmesartan 20 mg plus amlodipine 10 mg followed by amlodipine 10 mg/valsartan 160 mg

ELIGIBILITY:
Inclusion Criteria for Core study:

* Male or female patients (>=18 years)
* Females must be either post-menopausal for one year, surgically sterile or using effective contraceptive methods
* Patients with essential hypertension (diastolic blood pressure >=100 mmHg and <110 mmHg)

Inclusion Criteria for Extension:

- Patients had to have a msSBP >= 140 mmHg and/or msDBP >= 90 mmHg at week 8 ie, end of core study.

Exclusion Criteria for Core study:

* Severe hypertension (diastolic blood pressure >=110 mmHg or systolic blood pressure >= 180 mmHg)
* Pregnant or nursing women
* Treated hypertensive patients with controlled hypertension under current therapy
* A history of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, and heart failure NYHA II - IV

Exclusion Criteria for Extension:

* prematurely discontinued the core study
* failed to comply with the core study protocol

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Sponsor GmbH
Locations (2):
- Novartis Investigative Site, , Germany, Schwerin, Germany
- 30 sites in Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlodipine(AML)+Olmesartan, AML+Valsartan, AML+Valsartan+HCTZ: During the Treatment Phase 1, participants received 1 week of treatment with olmesartan 10 mg and amlodipine 5 mg once daily in free combination, followed by three weeks of treatment with olmesartan 20 mg plus amlodipine 10 mg once daily in free combination. During the Treatment Phase 2 participants received amlodipine 10 mg plus valsartan 160 mg for 4 weeks. During the Extension Phase, participants received 4 weeks treatment with amlodipine 10 mg plus valsartan 160 mg plus hydrochlorothiazide (HCTZ) 12.5 mg.
Period: Phase 1 - Amlodipine+Olmesartan
Arm/Group | Amlodipine(AML)+Olmesartan, AML+Valsartan, AML+Valsartan+HCTZ
Started | 257
Completed | 251
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Administrative problems | 1
Period: Phase 2 - Amlodipine+Valsartan
Arm/Group | Amlodipine(AML)+Olmesartan, AML+Valsartan, AML+Valsartan+HCTZ
Started | 176 (Only patients with mean sitting diastolic BP ≥ 90 mmHg at the end of Phase 1 entered this phase.)
Completed | 173
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Period: Phase 3 - Amlodipine+Valsartan+HCTZ
Arm/Group | Amlodipine(AML)+Olmesartan, AML+Valsartan, AML+Valsartan+HCTZ
Started | 91 (Only patients with systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg at the end of Phase 2.)
Completed | 91
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amlodipine(AML)+Olmesartan, AML+Valsartan, AML+Valsartan+HCTZ
Number analyzed (Participants) | 257
Age, Continuous [Mean (Standard Deviation); unit: years]
  Phase 1 - Amlodipine+olmesartan | 58.8 (12.38)
  Phase 2 - Amlodipine+valsartan | 59.8 (11.84)
  Phase 3 - Amlodipine+valsartan+HCTZ | 60.9 (10.98)
Sex/Gender, Customized [Number; unit: participants]
  Phase 1 - Amlodipine+olmesartan - Female | 112
  Phase 1 - Amlodipine+olmesartan - Male | 145
  Phase 2 - Amlodipine+valsartan - Female | 76
  Phase 2 - Amlodipine+valsartan - Male | 100
  Phase 3 - Amlodipine+valsartan+HCTZ - Female | 32
  Phase 3 - Amlodipine+valsartan+HCTZ - Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) During the Core Phase of the Study
Description: The arm in which the highest sitting diastolic pressures were found at study entry was the arm used for all subsequent readings. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, systolic/diastolic blood pressure were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements. A negative change indicates improvement.
Time Frame: Baseline Phase 2 (Week 4) to end of Phase 2 (Week 8)
Population: Intent-to-treat population (ITT): All patients who took at least one dose of amlodipine plus valsartan who had at least one primary efficacy parameter evaluation. Patients who dropped out were included in the ITT population if there was any BP measurement available; their last available blood pressure measurement was used for the analysis.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Amlodipine+Valsartan - Phase 2: Patients with uncontrolled mean sitting diastolic BP (msDBP ≥ 90 mmHg) at the end of Phase 1 were treated for 4 weeks with amlodipine 10 mg plus valsartan 160 mg taken orally in the morning.
Arm/Group | Amlodipine+Valsartan - Phase 2
Number analyzed (Participants) | 175
mmHg | -9.13 (1.97) [-10.19 to -8.06]

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) During the Core Phase of the Study
Description: as for outcome 1
Time Frame: Baseline Phase 2 (Week 4) to end of Phase 2 (Week 8)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine+Valsartan - Phase 2
Number analyzed (Participants) | 175
mmHg | -7.87 (9.48) [-9.33 to -6.11]

3. Secondary Outcome: Change in Sitting Pulse Pressure During the Core Phase of the Study
Description: Pulse pressure is systolic pressure (SP) minus diastolic pressure (DP). The arm in which the highest sitting DPs were found at study entry was the arm used for all subsequent readings. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, SP and DP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements. A negative change indicates improvement.
Time Frame: Baseline Phase 2 (Week 4) to end of Phase 2 (Week 8)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine+Valsartan - Phase 2
Number analyzed (Participants) | 175
mmHg | 1.26 (9.64) [0.49 to 3.01]

4. Secondary Outcome: Change in Sitting Pulse Rate During the Core Phase of the Study
Description: Pulse rate was measured once for 30 seconds just prior to blood pressure measurements in the sitting position.
Time Frame: Baseline Phase 2 (Week 4) to end of Phase 2 (Week 8)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: BPM (beats per minute)
Arm/Group | Amlodipine+Valsartan - Phase 2
Number analyzed (Participants) | 175
BPM (beats per minute) | -1.93 [-3.06 to -0.79]

5. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) During the Extension Phase of the Study
Description: as for outcome 1
Time Frame: Baseline Phase 3 (Week 8) to end of Phase 3 (Week 12)
Population: Safety population: All patients who took at least one dose of amlodipine 10 mg plus valsartan 160 mg plus HCTZ 12.5 mg.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Amlodipine+Valsartan+HCTZ - Phase 3: Patients with uncontrolled mean sitting systolic or diastolic blood pressure (msDBP ≥ 90 mmHg and/or msSBP ≥ 140 mmHg) at the end of Phase 2 were offered a 4 week treatment extension with amlodipine 10 mg plus valsartan 160 mg plus hydrochlorothiazide (HCTZ) 12.5 mg taken orally in the morning.
Arm/Group | Amlodipine+Valsartan+HCTZ - Phase 3
Number analyzed (Participants) | 91
mmHg | -5.22 [-6.76 to -3.68]

6. Secondary Outcome: Percentage of Patients Who Achieved Normalized Blood Pressure During the Core Phase of the Study
Description: Normalized Blood Pressure was defined as a msSBP < 140 mmHg and/or a msDBP < 90 mmHg.
Time Frame: Baseline Phase 2 (Week 4) to end of Phase 2 (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Amlodipine+Valsartan - Phase 2
Number analyzed (Participants) | 175
Percentage of participants
  msSBP < 140 mmHg | 44.6
  msDBP < 90 mmHg | 72.6

7. Secondary Outcome: Percentage of Patients Who Achieved a Protocol-defined Blood Pressure Response During the Core Phase of the Study
Description: Blood pressure response was defined as msSBP < 140 mmHg or a 20 mmHg decrease in msSBP at the end of Phase 2 (Week 8) compared to Baseline in Phase 2 (week 4) or a msDBP < 90 mmHg or a 10 mmHg decrease in msDBP at the end of Phase 2 compared to Baseline in Phase 2.
Time Frame: Baseline of Phase 2 (Week 4) to end of Phase 2 (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Amlodipine+Valsartan - Phase 2
Number analyzed (Participants) | 175
Percentage of participants
  msSBP response | 47.4
  msDBP response | 73.1

8. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) During the Extension Phase of the Study
Description: as for outcome 1
Time Frame: Baseline Phase 3 (Week 8) to end of Phase 3 (Week 12)
Population: Safety population: All patients who took at least one dose of amlodipine 10 mg plus valsartan 160 mg plus HCTZ 12.5 mg.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine+Valsartan+HCTZ - Phase 3
Number analyzed (Participants) | 91
mmHg | -10.84 [-12.94 to -8.75]

9. Secondary Outcome: Change in Sitting Pulse Pressure During the Extension Phase of the Study
Description: as for outcome 3
Time Frame: Baseline Phase 3 (Week 8) to end of Phase 3 (Week 12)
Population: Safety population: All patients who took at least one dose of amlodipine 10 mg plus valsartan 160 mg plus HCTZ 12.5 mg.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine+Valsartan+HCTZ - Phase 3
Number analyzed (Participants) | 91
mmHg | -5.62 [-7.74 to -3.50]

10. Secondary Outcome: Change in Sitting Pulse Rate During the Extension Phase of the Study
Description: Pulse rate was measured once for 30 seconds just prior to blood pressure measurements in the sitting position.
Time Frame: Baseline Phase 3 (Week 8) to end of Phase 3 (week 12)
Population: Safety population: All patients who took at least one dose of amlodipine 10 mg plus valsartan 160 mg plus HCTZ 12.5 mg.
Measure: Mean (95% Confidence Interval); unit: BPM (beats per minute)
Arm/Group | Amlodipine+Valsartan+HCTZ - Phase 3
Number analyzed (Participants) | 91
BPM (beats per minute) | 0.09 [-1.36 to 1.54]

11. Secondary Outcome: Percentage of Patients Who Achieved Normalized Blood Pressure During the Extension Phase of the Study
Description: Normalized Blood Pressure was defined as a msSBP < 140 mmHg and/or a msDBP < 90 mmHg.
Time Frame: Baseline Phase 3 (Week 8) to end of Phase 3 (Week 12)
Population: Safety population: All patients who took at least one dose of amlodipine 10 mg plus valsartan 160 mg plus HCTZ 12.5 mg.
Measure: Number; unit: Percentage of participants
Arm/Group | Amlodipine+Valsartan+HCTZ - Phase 3
Number analyzed (Participants) | 91
Percentage of participants
  msSBP < 140 mmHg | 59.3
  msDBP < 90 mmHg | 83.5

12. Secondary Outcome: Percentage of Patients Who Achieved a Protocol-defined Blood Pressure Response During the Extension Phase of the Study
Description: Blood pressure response was defined as msSBP < 140 mmHg or a 20 mmHg decrease in msSBP at the end of Phase 3 compared to Baseline in Phase 3 or a msDBP < 90 mmHg or a 10 mmHg decrease in msDBP at the end of Phase 3 compared to Baseline in Phase 3.
Time Frame: Baseline of Phase 3 (Week 8) to end of Phase 3 (Week 12)
Population: Safety population: All patients who took at least one dose of amlodipine 10 mg plus valsartan 160 mg plus HCTZ 12.5 mg.
Measure: Number; unit: Percentage of participants
Arm/Group | Amlodipine+Valsartan+HCTZ - Phase 3
Number analyzed (Participants) | 91
Percentage of participants
  msSBP response | 61.5
  msDBP response | 83.5

ADVERSE EVENTS:
Groups:
- Phase 1 - Amlodipine+Olmesartan: 4 weeks treatment with amlodipine 10 mg plus olmesartan 20 mg taken orally once daily in the morning.
- Phase 2 - Amlodipine+Valsartan: Patients with uncontrolled mean sitting diastolic BP (msDBP ≥ 90 mmHg) at the end of Phase 1 were treated for 4 weeks with amlodipine 10 mg plus valsartan 160 mg taken orally in the morning.
- Phase 3 - Amlodipine+Valsartan+HCTZ: Patients with uncontrolled mean sitting systolic or diastolic blood pressure (msDBP ≥ 90 mmHg and/or msSBP ≥ 140 mmHg) at the end of Phase 2 were offered a 4 week treatment extension with amlodipine 10 mg plus valsartan 160 mg plus hydrochlorothiazide (HCTZ) 12.5 mg taken orally in the morning.
Arm/Group | Phase 1 - Amlodipine+Olmesartan | Phase 2 - Amlodipine+Valsartan | Phase 3 - Amlodipine+Valsartan+HCTZ
Serious Adverse Events (participants affected / at risk) | 1/257 | 0/176 | 0/91
Other Adverse Events (participants affected / at risk) | 0/257 | 0/176 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Amlodipine+Olmesartan (N=257) | Phase 2 - Amlodipine+Valsartan (N=176) | Phase 3 - Amlodipine+Valsartan+HCTZ (N=91)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.